CLINICAL TRIAL: NCT04820192
Title: Effects of CranioSacral Therapy Upon Symptoms of Post-Acute Concussion and Post-Concussion Syndrome
Brief Title: Craniosacral Therapy for Concussion Symptoms
Status: Completed | Type: Observational
Sponsor: Special Therapies, Inc. (Other)
Responsible Party: Principal Investigator, Susan Vaughan Kratz, Clinical Director, Special Therapies, Inc.
Other Study IDs: CST for PCS
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Post-Concussion Syndrome
MeSH Terms: conditions — Post-Concussion Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Post-acute concussion (<6 months) or Post-Concussion Syndrome (PCS) (≥ 6 months): Patients were divided into cohort groupings to compare outcomes of applying CranioSacral Therapy to their unique constellations of persistent symptoms attributed to their concussion injury. Symptoms less than 3-6 months duration may be part of the usually rate of injury resolution through rest along. Symptoms persisting after 6 months are considered PCS. Less than 6 months since injury were considered post-acute concussion stage of recovery.
  Interventions: Other: Craniosacral Therapy
- Athletes (A) or Non-athletes (NA): Reporting of symptoms that exist and/or persist may differ between patients who are/were athletes and concussions were sustained during their sporting events. Non-athletes may report differently. The types of injuries involved in the concussion were also captured.
  Interventions: Other: Craniosacral Therapy
- Traditional gender.: Symptoms and response to rest has been reported to have differences between male and female patients. Age under 14 years was considered an exclusion due to immaturity in insight and reporting. Thus, young adult ages and older were included and observations between gender reporting was noted.
  Interventions: Other: Craniosacral Therapy

INTERVENTIONS:
Other: Craniosacral Therapy — The Upledger method of applying both specific and non-specific manual therapy of gentle, sustained, non-invasive stretch to soft tissues of fascia, meninges and osseous attachments. Fluid exchange is also believed to be a resulting result of CST. Treatment is applied to myofascial and osseous sites over the entire body, tending to specific and unique constellation of tissue restrictions and osseous compressions of soft tissue.

SUMMARY:
This study investigated the utilization of CranioSacral Therapy (CST) in patients with Post-Concussion Syndrome (PCS) and capture patient-reported perceptions of their lived experiences of treatment effect upon their symptoms. The first part part was a 10 year chart review of patients who sought out CST to capture data from the medical records. The second part was an anonymous post treatment survey.

ELIGIBILITY:
Inclusion Criteria:

* Charts were extracted from a group of 212 of patients with a history of concussion to a final chart review size of 67. These patients had specifically sought of CST to address symptoms of Post Concussion Syndrome.

Exclusion Criteria:

* Was determined for the 2nd part of study: Post Treatment Outcome Survey. Final group size of 47 excluded those under age 14 and those with confounding medical or personal issues or involved in litigation.

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Ten year retrospective chart review of patients who received craniosacral therapy addressing symptoms post concussion
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Patient-directed Utilization of CST | Through study completion. 1 year - study is now completed
  Data extracted from medical chart to study how many sessions patients participated in (addressing their presenting symptoms). Number of sessions were recorded.

SECONDARY OUTCOMES:
Demographic information | 3 months
  Additional data extracted from chart review to study trends of population sample included: gender differences in reporting, athletes/non-athletes reporting, time since injury, etiology of concussion (sports vs. non-sports).
Post-treatment Patient-reported Outcome Survey | Through study completion. 1 year - study is now completed
  Anonymous 10 question survey for participants meeting inclusion criteria from the original 67 (from chart review) recruited to complete an anonymous electronic survey. This survey highlighted symptoms they experienced from their concussions and if CST had any effect on any of the symptoms. Symptom list was extracted from the standard Post Concussion Symptom Checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Kratz, OTR, Principal Investigator — Special Therapies, Inc.
Locations (1):
- Special Therapies, Inc., Waukesha, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided